CLINICAL TRIAL: NCT06440759
Title: Evaluation of Efficacy and Safety Using oXiris Versus M100 Filter in Pneumonia-induced Acute Kidney Injury (AKI) Patients Requiring Continuous Renal Replacement Therapy (CRRT)
Brief Title: To Compare the Efficacy and Safety of Using oXiris and M100 During CRRT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mohd Zulfakar Mazlan, MBBS (Other)
Responsible Party: Sponsor-Investigator, Mohd Zulfakar Mazlan, MBBS, Associate Professor, Universiti Sains Malaysia
Organization: Universiti Sains Malaysia (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: USM/JEPeM/KK/23090718
Record Dates: First submitted 2024-04-30; First posted 2024-06-04 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: AKI - Acute Kidney Injury; Pneumonia
MeSH Terms: conditions — Acute Kidney Injury; Pneumonia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: single-blinding (patient)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- oXiris filter (Experimental): Continuous Renal Replacement Therapy with the adsorption membrane filter Oxiris.
  The specific septic biomarkers such as interleukin 6(IL-6), procalcitonin (PCT), C-reactive protein (CRP) along with other routine blood investigation results taken at the beginning of therapy and 24 hours after the treatment will be compared.
  The 28-day mortality will be recorded following treatment.
  Interventions: Device: oXiris filter
- M100 filter (Active Comparator): Continuous Renal Replacement Therapy with the adsorption membrane filter M100. The specific septic biomarkers such as interleukin 6(IL-6), procalcitonin (PCT), C-reactive protein (CRP) along with other routine blood investigation results taken at the beginning of therapy and 24 hours after the treatment will be compared.
  The 28-day mortality will be recorded following treatment.
  Interventions: Device: M100 filter

INTERVENTIONS:
Device: oXiris filter — Continuous Renal Replacement Therapy with the adsorption membrane filter Oxiris.
  The specific septic biomarkers such as interleukin 6(IL-6), procalcitonin (PCT), C-reactive protein (CRP) along with other routine blood investigation results taken at the beginning of therapy and 24 hours after the treatment will be compared.
  Arms: oXiris filter
Device: M100 filter — Continuous Renal Replacement Therapy with the adsorption membrane filter M100. The specific septic biomarkers such as interleukin 6(IL-6), procalcitonin (PCT), C-reactive protein (CRP) along with other routine blood investigation results taken at the beginning of therapy and 24 hours after the treatment will be compared.
  Arms: M100 filter

SUMMARY:
The purpose of this study aimed to compare the efficacy of Oxiris (Baxter) and M100 filters on IL-6 as primary outcomes and other blood cell counts, blood biochemistry (serum urea, creatinine, potassium, sodium), inflammation indicators (CRP, PCT), as secondary outcomes and safety (28 days mortality as a primary outcome and coagulopathy, lifespan of filter, usage of vasopressor, clinical conditions (ventilator-free days, ICU and hospital- length of stay) as a secondary outcome), clinical conditions (ventilator-free days, ICU and hospital- length of stay), and mortality of patients with pneumonia-related AKI.

DETAILED DESCRIPTION:
The type of hemofilter will be decided using a simple randomization. For the intervention group, only the oxiris filter will be used during the treatment period, while for the control group, the M100 filter will be used throughout the treatment. If the filter becomes clogged within 24 hours, the investigator will replace it with the same filter as the previous one. However, if the filter becomes clogged after 24 hours and the patient still requires CRRT, the investigator will replace it with M100. This change in filter type will not affect the study results, as only the blood parameters during the first 24 hours of treatment will be evaluated for objective one. The oxiris filter will be used for the first 24 hours, or whichever is longer, and will be replaced with an M100 filter if indicated for both groups. Therefore, it will not affect the outcome of objective two compared to the standard arm group

Termination of CRRT will be done according to recent studies once the patient fulfills either one or more of these criteria: urine output and serum creatinine are indicative of kidney recovery, vasopressor cessation, increased urine output ≥500ml/24H without diuretics, correction of fluid overload, hemodynamic stability and the possible need to shift to intermittent dialysis.

The patient will be followed up until 28 days following ICU admission. To avoid any missing data, at least 3 contact numbers will be made available. If unable to get in contact with the patient, the application status of alive or dead will be applied to a national registry.

ELIGIBILITY:
Inclusion Criteria:

* All adult patients aged>18 years old
* Diagnosis of septic shock
* Diagnosis of KDIGO stage 3 acute renal failure

Exclusion Criteria:

* Moribund patient or patient that is expected to die within 72 hours
* Pregnancy
* patient with a bleeding tendency or known allergy to heparin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-05-30 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
To measure the effectiveness of the oxiris filter in reducing septic biomarker levels IL-6 | 24 hours
  To measure the effectiveness of oxiris filter compared to the M100 filter in reducing the septic biomarker levels during CRRT. The baseline IL6 will be measured immediately before CRRT and post-CRRT
To compare the 28-days mortality of using oxiris filter during CRRT | 28 days
  To measure the 28-day mortality rate when using oxiris and M100 filter for CRRT. The 28-day mortality rate is calculated based on the number of deaths occurring within 28 days from a defined starting point, the start of CRRT.

SECONDARY OUTCOMES:
To compare the risk infection of by using oxiris during CRRT | 28 days
  To measure the risk of infection rate when using oxiris filter for CRRT. An infection is defined as an infection of the CRRT catheter such as CRBSI.
To compare the risk bleeding of using oxiris during CRRT | 28 days
  To measure the risk of bleeding rate when using oxiris filter for CRRT. Bleeding is defined as any bleeding noted such as gastrointestinal, urinary bleeding or respiratory tract bleeding.
To compare the risk of ventilator-free days of using oxiris during CRRT | 28 days
  To measure the risk of ventilator-free day rate when using oxiris filter for CRRT. It is defined as the number of days within a specific period (usually 28 days) during which a patient is both alive and free from mechanical ventilation. For example, if a patient is on mechanical ventilation for 10 days and survives the entire 28-day period, they would have 18 ventilator-free days (28 - 10 = 18). If a patient dies at any point within the 28 days, their VFDs would be zero.
To measure the effectiveness of the oxiris filter in reducing septic biomarker levels PCT | 24 hours
  To measure the effectiveness of oxiris filter compared to the M100 filter in reducing the septic biomarker levels during CRRT. The baseline PCT will be measured immediately before CRRT and post-CRRT
To measure the effectiveness of the oxiris filter in reducing septic biomarker levels CRP | 24 hours
  To measure the effectiveness of oxiris filter compared to the M100 filter in reducing the septic biomarker levels during CRRT. The baseline CRP will be measured immediately before CRRT and Post CRRT

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universiti Sains Malaysia (HUSM), Kubang Kerian, Kelantan, Malaysia